CLINICAL TRIAL: NCT01203410
Title: BilirubinProduction in Healthy Term Infants as Measured by Carbon Monoxide in Breath
Brief Title: Prediction of Jaundice in Term Infants
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Responsible Party: David K. Stevenson/ Lead Principal Investigator, Stanford University
Other Study IDs: NICHD-NRN-0004; U10HD021364 (NIH); U10HD027853 (NIH); U10HD027851 (NIH); U01HD019897 (NIH); U10HD027856 (NIH); U10HD027881 (NIH); U10HD027880 (NIH); U10HD021415 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027904 (NIH); U10HD027871 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Jaundice
Keywords: NICHD Neonatal Research Network; Term infant; Hyperbilirubinemia
MeSH Terms: conditions — Jaundice; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Term infants >2500g birthweight.

SUMMARY:
The objective of this study was to describe total bilirubin production in healthy term infants as a means of understanding the differences in jaundice pigment production associated with various common clinical circumstances.

DETAILED DESCRIPTION:
Jaundice occurs in most human neonates during the several days after birth. The objective of this study was to describe total bilirubin production in healthy term infants as a means of understanding the differences in jaundice pigment production associated with various common clinical circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Infants born via cesarean delivery (to ensure subjects would still be hospitalized and available for ETCOc measurement and blood sampling on day 3 postpartum)
* Delivery within each center's scheduled recruitment period (to maximize nursing availability and minimize cost)
* Birth weight >2500 g
* Gestational age >37 weeks

Exclusion Criteria:

* Any illness that would require admission to the neonatal intensive-care unit (NICU) within 8 hours of birth

Max Age: 8 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term infants.
Sampling Method: Probability Sample
Enrollment: 535 (Actual)
Dates: Start 1991-11; Primary Completion 1992-11 (Actual); Study Completion 1992-11 (Actual)

PRIMARY OUTCOMES:
End-tidal carbon End-tidal carbon monoxide levels corrected for ambient air (ETCOc) | 2-8 hours of age
  An index of bilirubin production

CONTACTS AND LOCATIONS:
Overall Officials: David K. Stevenson, MD, Study Director — Stanford University; William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University; James A. Lemons, MD, Principal Investigator — Indiana University; Raymond Bain, PhD, Principal Investigator — George Washington University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Jon E. Tyson, MD, Principal Investigator — University of Texas; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Charles R. Bauer, MD, Principal Investigator — University of Miami; Barbara J. Stoll, MD, Principal Investigator — Emory University; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (13):
- United States (13):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] Vreman HJ, Stevenson DK, Oh W, Fanaroff AA, Wright LL, Lemons JA, Wright E, Shankaran S, Tyson JE, Korones SB, et al. Semiportable electrochemical instrument for determining carbon monoxide in breath. Clin Chem. 1994 Oct;40(10):1927-33. PMID 7923774
- [Result] Stevenson DK, Vreman HJ, Oh W, Fanaroff AA, Wright LL, Lemons JA, Verter J, Shankaran S, Tyson JE, Korones SB, et al. Bilirubin production in healthy term infants as measured by carbon monoxide in breath. Clin Chem. 1994 Oct;40(10):1934-9. PMID 7923775
- [Result] Vreman HJ, Verter J, Oh W, Fanaroff AA, Wright LL, Lemons JA, Shankaran S, Tyson JE, Korones SB, Bauer CR, Stoll BJ, Papile LA, Donovan EF, Ehrenkranz RA, Stevenson DK. Interlaboratory variability of bilirubin measurements. Clin Chem. 1996 Jun;42(6 Pt 1):869-73. PMID 8665677
- [Result] Hintz SR, Gaylord TD, Oh W, Fanaroff AA, Mele L, Stevenson DK, Nichd FT; NICHD, Neonatal Research Network. Serum bilirubin levels at 72 hours by selected characteristics in breastfed and formula-fed term infants delivered by cesarean section. Acta Paediatr. 2001 Jul;90(7):776-81. PMID 11519981
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/